CLINICAL TRIAL: NCT02494284
Title: Short-Term Dual Antiplatelet and Maintenance CloPidogrel Therapy After Drug-Eluting Stent Implantation : STAMP-DES Trial
Brief Title: Short-Term Dual Antiplatelet and Maintenance CloPidogrel Therapy After Drug-Eluting Stent Implantation
Acronym: STAMP-DES
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: CHEOL WHAN LEE, M.D., Ph.D (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Medtronic (Industry); Chong Kun Dang Pharmaceutical Corp. (Industry)
Responsible Party: Sponsor-Investigator, CHEOL WHAN LEE, M.D., Ph.D, M.D., Ph,D, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2014-09
Record Dates: First submitted 2015-07-05; First posted 2015-07-10 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Dual antiplatelet platelet therapy; Drug eluting stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short term dual therapy (Experimental)
  Interventions: Drug: Clopidogrel
- Long term dual therapy (Active Comparator)
  Interventions: Drug: Aspirin plus clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — 6-month DAPT followed by clopidogrel monotherapy
  Arms: Short term dual therapy
Drug: Aspirin plus clopidogrel — standard long-term dual antiplatelet strategies (24-month DAPT followed by aspirin monotherapy)
  Arms: Long term dual therapy

SUMMARY:
The purpose of this study is to compare short-term (6-month Dual Anti Platelet Therapy(DAPT) followed by clopidogrel monotherapy) vs. standard long-term dual antiplatelet strategies (24-month DAPT followed by aspirin monotherapy) on clinically relevant bleeding complications (Bleeding Academic Research Consortium(BARC) type 2, 3, or 5)31 in patients after zotarolimus-eluting stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 19 years of age
* Patients with stable coronary artery disease who were successfully treated with zotarolimus-eluting stents
* Patients without major bleeding or MACE (myocardial infarction, stent thrombosis, stoke, repeat revascularization) within 6 months after zotarolimus-eluting stent placement
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Persistent thrombocytopenia (platelet count <100,000/µl)
* A known intolerance to a study drug (aspirin, clopidogrel)
* Patients requiring long-term oral anticoagulants or cilostazol
* Patients presented with acute myocardial infarction (STEMI or NSTEMI) at the time of index procedure
* Planned cardiac surgery (e.g., CABG, valve repair or replacement, or aneurysmectomy) or planned major non-cardiac surgery within 18 months after procedure
* Bare-metal stent implantation at the time of index procedure
* Chronic disease requiring treatment with oral, intravenous, or intra-articular corticosteroids (use of topical, inhaled, or nasal corticosteroids is permissible).
* A diagnosis of cancer in the past 2 years or current treatment for the active cancer.
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
* Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 3 times upper limit of normal).
* History of adult asthma manifested by bronchospasm in the past 6 months, or currently taking regular anti-asthmatic medication(s).
* Unwillingness or inability to comply with the procedures described in this protocol.
* Patients pregnant or breast-feeding or child-bearing potential.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinically relevant bleeding | 18 months
  clinically relevant bleeding (Bleeding Academic Research Consortium Definition: type 2, 3, or 5) at 18 months after randomization (6-24 months after the procedure)

SECONDARY OUTCOMES:
Number of participants with death from cardiovascular cause | 18 months
Number of participants with myocardial infarction | 18 months
Number of participants with stroke | 18 months
Number of participants with stent thrombosis | 18 months
Number of participants with repeat revascularization | 18 months
Number of participants with BARC(Bleeding Academic Research Consortium Definition) type 3 or 5 | 18 months
Number of participants with a composite of death from vascular causes or myocardial infarction | 18 months
Number of participants with a composite of death from cardiovascular causes, myocardial infarction, stroke, stent thrombosis | 18 months
Number of participants with a composite of death from vascular causes, myocardial infarction, stroke, stent thrombosis, BARC type 3 or 5 | 18 months
Number of participants with gastrointestinal side effects (gastric or duodenal active ulcer, perforation, gastrointestinal bleeding) | 18 months
Number of participants with a composite of BARC(Bleeding Academic Research Consortium Definition) 2, 3, 5 or gastrointestinal side effects. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, Principal Investigator — Asan Medical Center; Cheol-Whan Lee, MD, Principal Investigator — Asan Medical Center
Locations (12):
- South Korea (12):
  - Keimyung University Dongsan Medical Center, Daegu
  - Eulji University Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Inje University Ilsan Paik Hospital, Ilsan
  - Cheju Halla General Hospital, Jeju City
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - Kyunghee University Medical Center, Seoul
  - SMA-SNU Boramae Medical Center, Seoul
  - The Catholic University of Korea St. Paul's Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan